CLINICAL TRIAL: NCT02233387
Title: Non Invasive Imaging of [18F]HX4 With Positron-Emission-Tomography (PET) in Cervix Cancer.
Brief Title: PET CT With HX4 in Cervix Cancer
Acronym: HX4-cervix
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: patients did not want to participate
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-36-14/12
Record Dates: First submitted 2012-02-29; First posted 2014-09-08 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Cervix Cancer
Keywords: cervix cancer; [18F] HX4 PET imaging; hypoxia; phase II trial
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypoxia | interventions — Injections; Magnetic Resonance Spectroscopy; 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F] HX4 PET imaging (Experimental): injection with [18F] HX4 and PET imaging at baseline and after 20 Gy radiotherapy
  Interventions: Other: injection with [18F] HX4 and PET imaging

INTERVENTIONS:
Other: injection with [18F] HX4 and PET imaging — A standard clinical [18F]FDG PET-CT will be performed for the radiotherapy planning.
  After a minimum time interval of 24 hours, baseline [18F]HX4 PET scans will be performed:
  Based on the phase I trial1 444 MBq (12 mCi) [18F]HX4 is administrated via a bolus IV injection.
  The first image acquisition is started together with the administration of [18F]HX4 (30-40 min dynamic). Static scans are acquired at 90 min, 180 min and 240 min p.i
  Other Names: 3-[18F]fluoro- 2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1- yl)propan-1-ol

SUMMARY:
The aim of this study is:

1. to determine if tumor hypoxia can be accurately visualised with [18F]HX4 PET imaging in cervix cancer,
2. to correlate the [18F]HX4 PET images with blood and tissue markers,
3. to investigate the quality and optimal timing of [18F]HX4 PET images,
4. to compare [18F]HX4 PET uptake with [18F]FDG PET uptake before and after treatment and
5. analyze correlation with responses

DETAILED DESCRIPTION:
Tumor hypoxia is the situation where tumor cells are or have been deprived of oxygen. Hypoxic tumor cells are usually more resistant to radiotherapy and chemotherapy and more likely to develop metastasis. In Cervix cancer, tumor hypoxia is known to be an important prognostic factor for long term survival. [18F]HX4 is being developed as a diagnostic radiopharmaceutical for PET imaging to find a marker for hypoxia that can be used in standard clinical practice. Current hypoxia tracers lack reliable image quality and kinetics. Because of the short half life and clearance, the investigators expect that [18F]HX4 will have a higher tumor to background ratio than current nitro-imidazole hypoxia markers such as [18F]-misonidazole. In a recent phase 1 clinical study from van Loon et al, PET-imaging with [18F]HX4 was feasible without any toxicity. The clinical use of a reliable, non-invasive and easy to use hypoxia imaging agent could allow selection of patients most likely to benefit from hypoxia modifying therapies.

ELIGIBILITY:
Inclusion criteria

* Histologically confirmed cervix carcinoma (squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma)
* tumor stages FIGO IB - IVA
* WHO performance status 0 to 2
* Scheduled for primary curative radiotherapy (either or not combined with chemotherapy or hyperthermia)
* No previous surgery to the Cervix
* No previous radiation to the Cervix
* The patient is willing and capable to comply with study procedures
* 18 years or older
* Written informed consent before patient registration

Exclusion criteria

* Recent (< 3 months) myocardial infarction
* Uncontrolled infectious disease
* Pregnant or breast feeding and/or not willing to take adequate contraceptive measures during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Visualisation of tumor hypoxia with [18F] HX4 PET imaging | 2 year
  Visualisation of tumor hypoxia with [18F] HX4 PET imaging

SECONDARY OUTCOMES:
Observation of spatial and temporal stability of [18F] HX4 PET images | 2 year
  Observation of spatial and temporal stability of [18F] HX4 PET images
Correlations with Complete Remission rates at 3 months restaging evaluation | 2 year
  Correlations with Complete Remission rates at 3 months restaging evaluation
Image quality of [18F] HX4-PET at different time points | 2 year
  Image quality of [18F] HX4-PET at different time points
Kinetic analysis of HX4 | 2 year
  Kinetic analysis of HX4
Correlation of hypoxia imaging with blood hypoxia markers (osteopontin, circulating CA-IX) | 2 year
  Correlation of hypoxia imaging with blood hypoxia markers (osteopontin, circulating CA-IX)
Correlation of hypoxia imaging with tumor tissue biomarkers (HPV, CA-IX, VEGF, EGFR, CD44, HIF-1α, mir-210) and autophagy related genes | 2 year
  Correlation of hypoxia imaging with tumor tissue biomarkers (HPV, CA-IX, VEGF, EGFR, CD44, HIF-1α, mir-210) and autophagy related genes
Spatial correlation of [18F] HX4-PET with [18F] FDG PET pre-treatment | 2 year
  Spatial correlation of [18F] HX4-PET with [18F] FDG PET pre-treatment
Spatial correlation of [18F] HX4-PET with [18F] FDG PET three months after treatment | 2 year
  Spatial correlation of [18F] HX4-PET with [18F] FDG PET three months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, prof MD PhD, Study Director — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Netherlands